CLINICAL TRIAL: NCT05314244
Title: A Prospective Randomized Comparison Between Pylorus-resecting and Preserving Pancreaticoduodenectomy on Postoperative Delayed Gastric Emptying and Nutritional Status
Brief Title: Comparison Between Pylorus-resecting and Preserving Pancreaticoduodenectomy on Delayed Gastric Emptying and Nutrition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Song Cheol Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DGE_2022
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Pancreaticoduodenectomy; Delayed Gastric Emptying; Nutrition
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pylorus resecting group (Experimental): The patients who underwent pylorus resecting pancreaticoduodenectomy for periampullary tumors
  Interventions: Procedure: Pylorus resecting pancreaticoduodenectomy
- pylorus preserving group (No Intervention): The patients who underwent pylorus preserving pancreaticoduodenectomy for periampullary tumors

INTERVENTIONS:
Procedure: Pylorus resecting pancreaticoduodenectomy — The patients in pylorus resection group will underwent pylorus resecting procedure during pancreaticoduodenectomy
  Arms: pylorus resecting group

SUMMARY:
Pylorus preserving pancreaticoduodenectomy has been standard procedure for periampullary benign and malignant disease. Delayed gastric emptying is one of most common complications after the procedure. Recently, pylorus resecting pancreaticoduodenectomy has been actively performed because some studies reported that the procedure can reduce postoperative delayed gastric emptying.

However, the level of evidence is low and there was few studies considering nutritional status after pylorus resecting pancreaticoduodenectomy.

The purpose of this study is to compare between pylorus-resecting and preserving pancreaticoduodenectomy on postoperative delayed gastric emptying and nutritional status.

DETAILED DESCRIPTION:
Pylorus preserving pancreaticoduodenectomy has been standard procedure for periampullary benign and malignant disease. Delayed gastric emptying is one of most common complications after the procedure. It can lead to delay initiation of adjuvant chemotherapy as well as postoperative recovery. Since 2010, pylorus resecting pancreaticoduodenectomy was introduced to reduce postoperative delayed gastric emptying. The cases have been actively increased. However, several prospective randomized controlled trials reported pylorus resection during pancreaticoduodenectomy did not reduce the incidence or severity of delayed gastric emptying. Recent meta-analysis also showed same results.

Previous randomized controlled trials were single center studies participating a relatively small number of patients. A large-scale multicenter study is needed to obtain high level of evidence. And nutritional difference may appear between pylorus preservation and resection groups. Few studies have dealt with nutritional status between two groups.

* This study aimed to compare between pylorus-resecting and preserving pancreaticoduodenectomy on postoperative delayed gastric emptying and nutritional status in 5 tertiary referral centers in Korea..
* A case of pancreaticoduodenectomy with periampullary benign and malignant tumors will be included. The expected number of patients is 394. The pylorus resecting group was performed in the experimental group and the pylorus preserving group was performed in control group.

This clinical study is a randomized prospective comparative study of the outcome of pylorus resecting and preserving pancreatoduodenectomy, and the research hypothesis is as follows.

* Nursing Hypothesis: There is no difference in incidence of delayed gastric emptying between patients who underwent pylorus resecting pancreaticoduodenectomy and patients who underwent pylorus preserving surgery.
* Alternative Hypothesis: Based on the results of the same operation of the existing institution, the average incidence of delayed gastric emptying for pylorus preserving pancreaticoduodenectomy is estimated to be 20%, and the average incidence of delayed gastric emptying for pylorus resecting pancreaticoduodenectomy is estimated to be 10%.

The random assignment of this study is assigned according to the order of assignment in the planning stage of the study as a block randomization scheme with appropriate block size set.

* Plan for recruitment of research subjects : All patients scheduled for open pancreaticoduodenectomy for pancreatic or periampullary lesions will be explained about this study and will be selected after informed consent.
* Operative method : Both patients underwent conventional open pancreaticoduodenectomy with or without pylorus resection. In the experimental group, stomach resection was performed 1.0cm proximal to pylorus. In the control group, duodenal resection was performed 2.0cm distal to pylorus. Both groups are performed through the same surgical procedure except pylorus preservation or resection and the procedure is as follows. Kocher maneuver is performed to mobilize the duodenum. Omentectomy is performed and the gastrocolic truck is identified and ligated. The stomach or duodenum is cut off using an automatic stapler. A cholecystectomy is performed. The bile duct is cut and the frozen section is checked to confirm whether the tumor is invaded. The hepatic and hepatic arteries are dissected and the surrounding lymph nodes are dissected. The gastroduodenal artery is detached and ligated. The pancreas is cut from the pancreas neck, and the tumor is examined by freezing biopsy. The proximal plant is dissected and cut, and the pancreas uncinate process is released from the superior mesenteric artery and vein. Pancreaticojejunal anastomosis, hepaticojejunal anastomosis, gastrojejunal or duodenojejunal anastomosis are performed. In this case, anastomosis is performed by the method used by each institution.

Patient management after surgery

* preoperative : NRI(weight, albumin), BMI, Blood chemistry, Abdomen&Pelvic Computed Tomography(APCT) (body composition calculation)
* 1day after surgery : blood chemistry, removal of nasogastric tube, water intake, early gate
* 2days after surgery : start diet (liquid or solid)
* 3days after surgery : blood chemistry, intravenous patient controlled analgesia removal, after 3 days, considering drain amylase and drain volume it can be removed.
* 5days after surgery : APCT
* 7days after surgery : NRI(weight, albumin), blood chemistry, tumor marker(if pathology is malignant)
* 14days after surgery : NRI(weight, albumin), blood chemistry
* 21days after surgery : NRI(weight, albumin), blood chemistry
* 3months after surgery : NRI(weight, albumin), blood chemistry, APCT (body composition check)
* 6months after surgery : NRI(weight, albumin), blood chemistry, APCT (body composition check)
* 12months after surgery : NRI(weight, albumin), blood chemistry, APCT(body composition check)

  ** Daily check amount of food intake from operation to discharge(Grade 1~3)
* Grade I: 30% or less of the provided amount can be consumed
* Grade II: 30~50% of the provided amount can be consumed
* Grade III: 50% or more of the provided amount can be consumed

  * Nutritional risk index (NRI) was calculated using the following formula: NRI = (1.519 × serum albumin g/L) + 0.417 × (present weight/usual weight) × 100, with usual weight being the value measured during preoperative evaluation period

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 79 years
* Performance: Eastern Cooperative Oncology Group (ECOG) 0-2
* The preoperative examination showed that the lesion could invade to major artery.
* No distant metastasis
* Bone marrow function: white blood cell (WBC) at least 3,000 / mm3, Platelet count at least 100,000 / mm3
* Liver function : aspartate transaminase (AST)/alanine transaminase(ALT) less than 3 times upper limit of normal
* Kidney function: Creatinine no greater than 1.5 times upper limit of normal.
* Patients who consented to and signed the consent

Exclusion Criteria:

* Patients diagnosed with duodenal cancer
* Those with active or uncontrolled infections
* Those with severe psychiatric / neurological disorders
* Alcohol or other drug addicts
* Patients who underwent previous major abdominal surgery (ex. gastrectomy, colectomy)
* Patients included in other clinical studies that may affect this study
* Patients who cannot follow the directions of the researcher
* Those with uncontrolled heart disease
* Patients with moderate or severe comorbidities who are thought to have an impact on quality of life or nutritional status (ex. cirrhosis, chronic kidney failure, heart failure, etc.)
* Pelvic tumor, benign tumor, malignant tumor in other organs
* Patients who received prior chemotherapy
* In addition to the planned pancreaticoduodenectomy, patients who require resection of other major abdominal organs, such as gastrectomy, colectomy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 394 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2024-04-28 (Estimated); Study Completion 2025-04-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of delayed gastric emptying | up to 1 months
  Delayed gastric emptying(DGE) is defined by International Study Group of Pancreas Surgery(ISGPS) definition.
  * Grade A DGE should be considered if the Nasogastric tube(NGT) is required between the Postoperative Day(POD) 4 and 7, or if reinsertion of the NGT was necessary owing to nausea and vomiting after removal by POD 3 and the patient is unable to tolerate a solid diet on POD 7, but resumes a solid diet before Postoperative Day(POD)14 ** Grade B DGE is present if the NGT is required from POD 8-14, if reinsertion of the NGT was necessary after POD 7, or if the patient cannot tolerate unlimited oral intake by Postoperative Day(POD)14, but is able to resume a solid oral diet before POD 21 *** Grade C DGE is present when nasogastric intubation cannot be discontinued or has to be reinserted after POD 14, or if the patient is unable to maintain unlimited oral intake by POD 21

SECONDARY OUTCOMES:
Nutritional risk index(NRI) | up to 12 months
  Nutritional risk index (NRI) is calculated using the following formula: NRI = (1.519 × serum albumin g/L) + 0.417 × (present weight/usual weight) × 100, with usual weight being the value measured during preoperative evaluation period
Sarcopenia | up to 12 months
  Body composition, including Skeletal muscle area(SMA), Subcutaneous fat area(SFA), Visceral fat area(VFA) is calculated by axial CT slice at the L3 vertebral inferior endplate level

CONTACTS AND LOCATIONS:
Overall Officials: Song-Cheol Kim, MD-PhD, Principal Investigator — Asan Medical Center

IPD SHARING:
Plan to Share IPD: No